CLINICAL TRIAL: NCT02150811
Title: Longitudinal Change of Distribution Pattern of Hunner's Ulcer in Patient With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Observational Study of Hunner's Ulcer in Patient With Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Soo Choo, Professor, Asan Medical Center
Other Study IDs: 20131119
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hunner's ulcer

SUMMARY:
The purpose of this study is to observe change of distribution pattern of Hunner's ulcer in patient with interstitial cystitis/bladder pain syndrome

DETAILED DESCRIPTION:
This is observational, 12 months study

ELIGIBILITY:
Inclusion Criteria:

1. must have experienced bladder pain, urinary urgency and urinary frequency, for at least 6 months prior to entry into the study
2. Pain VAS ≥4
3. O'Leary-Sant Interstitial Cystitis questionnaire (IC-Q) symptom and problem ≥ 12( and pain ≥2, and nocturia ≥ 2)
4. PUF score ≥ 13
5. cystoscopic record within 2 years
6. Hunner ulcer lesion in cystoscopic finding

Exclusion Criteria:

1. Scheduled for or use of intravesical therapy (eg, bladder distention,transurethral resection of bladder ulcer, instillation) during or within 6months prior to the study and use of pentosan polysulfate sodium within 1 months prior to the study
2. Patients who are pregnancy or, childbearing age without no contraception
3. Patients with voided volume <40 or, > 400ml
4. Patients with microscopic hematuria, (≥1+ in dipstick), If not excluded that no evidence of neoplastic tumor examination
5. Patients with urine culture showing evidence of urinary tract infection 1month prior to the study
6. Accompanied medical problem below

   * Tuberculosis in urinary system
   * Bladder cancer, urethral cancer, prostate cancer
   * Recurrent cystitis
   * Anatomical disorder
7. Patients had prior surgery (eq, bladder augmentation, cystectomy
8. Patients with neurologic disorder
9. Patients with indwelling catheter or intermittent self-catheterization
10. Patients with psychologic problem

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Change of distribution pattern of Hunner's ulcer | 1 month, 6month, 12month

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No